CLINICAL TRIAL: NCT05346120
Title: Post-Acute COVID-19, Inflammation, and Depression
Acronym: COVID Long
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started
Sponsor: Sean Savitz (Other)
Responsible Party: Sponsor-Investigator, Sean Savitz, Neurologist, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID long
Record Dates: First submitted 2022-04-24; First posted 2022-04-26 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Post COVID -19 Depression

STUDY DESIGN:
Intervention Model Description: Single site, double blind, placebo-controlled, longitudinal study with a 1:1 ratio randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind for subject and investigator. Only unblinded is the Cellular Therapy Core which manufactures, randomizes and dispenses MSCs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Single IV infusion of 6 million cells/kg allogeneic marrow stromal cells (MSCs) lasting approximately 30 minutes
  Interventions: Biological: allogeneic marrow stromal cells (MSCs)
- Placebo controlled (Placebo Comparator): PlasmaLyte A supplemented with 5% HSA
  Interventions: Biological: allogeneic marrow stromal cells (MSCs)

INTERVENTIONS:
Biological: allogeneic marrow stromal cells (MSCs) — stem cell infusion

SUMMARY:
Single site, double blind, placebo-controlled, longitudinal study of depression in Subjects with COVID- 19 long haulers syndrome using a 1:1 ratio randomization for a single IV infusion of 6 million cells/kg allogeneic marrow stromal cells (MSCs).

DETAILED DESCRIPTION:
A prospective study evaluating depression in COVID- 19 long haulers syndrome treated with allogeneic marrow stromal cells. Accruing evidence suggests cognitive and affective dysfunction, depression, and fatigue occur after COVID-19 infection. These impairments, likely arise from multiple factors that may include cell/organ damage due to direct viral infection or inflammatory process. The current proposal hypothesizes that the inflammatory response is a critical mechanism underlying these neuropsychiatric conditions.

After recovery from COVID-19, the hyperimmune activity secondary to tissue damages and endothelial activation may leave post-acute COVID-19 patients vulnerable to the neural consequences of proinflammatory cytokines Heightened inflammation can alert the central nervous system to induce sickness behaviors and elevated risk of depression.

We hypothesize that allogeneic marrow stromal cells (MSCs) will attenuate post-covid inflammation and reduce the resulting neuropsychiatric symptoms.

Aim 1: Evaluate the feasibility and acceptability of recruiting, providing MSC/sham infusions, and following participants to collect biomarker and clinical outcomes.

• MSC's infusions, baseline and follow-up measurements will be feasible and acceptable to participants.

Aim 2: Estimate the probability of demonstrating improvement in depression (i.e. > 30% reduction on the MADRS) among adult patients experiencing post-COVID depression randomized to MSC Infusion versus Sham Infusion. To determine (obtain, evaluate, verify, etc.) …

• MSC Infusion will out-perform Sham Infusion on the proportion of MADRS responders.

Aim 3: Relative to usual care, estimate the differential improvement of MSC-treated participants on cognitive measures and PROMIS (Health-Related Quality of Life; HRQOL) scales (e.g. Fatigue, Pain, Anger, Anxiety, etc.).

• MSC Infusion will out-perform Sham Infusion +on improvements in cognitive function and HRQOL measures.

Aim 4: Estimate the change attributable to MSC treatment on a panel of inflammatory biomarkers relative to usual care.

• Relative to Sham Infusion, MSC Infusion will down-regulate pro-inflammatory processes while upregulating anti-inflammatory processes, and this modulation will be related to improvement in depression, cognitive and PROMIS measures. Relative to Sham Infusion, MSC Infusion will down-regulate pro-inflammatory processes while upregulating anti-inflammatory processes, and this modulation will be related to improvement in depression, cognitive, and PROMIS measures.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject, or legally authorized representative, must be able to understand and voluntarily sign an informed consent document 2. Diagnosed with COVID-19 within the last 90 days 3. Age 18 to 80 years 4. QIDS-SR> 11

Exclusion Criteria:

* 1. A pre-COVID-19 history of cognitive dysfunction, or chronic fatigue 2. Exclude Recurrent episodes of depression (allowed: a prior episode but completed medication at least 3 months before enrollment) 3. Any medical or psychiatric condition which could confound study assessments 4. Stroke within the last 3 months 5. Developmental delay 6. Any other condition that the investigator feels would pose a significant hazard to the patient if enrolled 7. Current participation in any interventional research study 8. Unable to return for follow-up visits for clinical evaluation, laboratory studies, or imaging evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology (QIDS-SR) | from pre-infusion to Day 90
  depression rating scale

SECONDARY OUTCOMES:
PROMIS | from pre-infusion to Day 90
  Health related quality of life and scales measuring fatigue, pain, anger, anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Alderman, PhD, Study Director — UTHealth Science Center Houston

IPD SHARING:
Plan to Share IPD: No